CLINICAL TRIAL: NCT04105894
Title: Does Gastric Reflux Induce Sinonasal Symptoms?
Brief Title: Gastric Reflux and Sinonasal Symptoms
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rehab Abdelale Mohammed, Resident in Otorhinolaryngology Department, Assiut University
Other Study IDs: GR & sinonasal symptoms
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Gastric Reflux; Gastro Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MSCT of nose and PNs — MSCT of nose and PNs axial, coronal and sagittal cuts without contrast to evaluate the state of the sinuses at the beginning of evaluation and after 2 months duration of medical treatment for GERD
Diagnostic Test: Swab from nasal and oral mucous discharge to evaluate presence of HCL and pepsin — Swab from nasal and oral mucous discharge to evaluate presence of HCL and pepsin at the at the beginning of evaluation and after 2 months duration of medical treatment for GERD
Drug: medical treatment of GERD t — medical treatment of GERD only for 2 months as described by gastroenterology department

SUMMARY:
The study is conducted to:

* study correlation between sinonasal troubles & GERD
* Assess whether antireflux therapy improve state of sinus in patients complaining from reflux & sinonasal symptoms

DETAILED DESCRIPTION:
Gatroesophageal reflux disease(GERD) is one of the most common diagnoses made by both primary care physicians and gastroenterologists . It is defined as a gastrointestinal motility disorder that results from the reflux of stomach contents into the esophagus or oral cavity, causing symptoms or complications .The prevalence of GERD is estimated to be between 20 and 30% of adults in western countries.

Some studies have found a correlation between GERD and certain diseases of the airway and a proposed association to others. Both asthma and laryngitis can be caused by GERD. Pepsin has been discovered in the middle ear of children with middle ear effusion and GERD has been implicated in the pathophysiology of otitis media with effusion. The authors conclude that there may be a role of antireflux therapy in patients with otitis media with effusion. The relationship between reflux and snoring/obstructive sleep apnea syndrome (OSAS) has been studied, and it is known that OSAS patients have a high incidence of nocturnal gatroesophageal reflux (nGER).

The coexistence of reflux and various respiratory disorders can be used to argue that there is probably a correlation between reflux and CRS. Though some data indicate an association between GERD and upper airway inflammatory disease, this remains a matter of controversy in today's medicine. It is suggested that, if an upper or lower respiratory tract disorder is causally related to GERD, certain criteria should be met:

1. An increased coexistence of both disorders should exist compared to the general population.
2. A biologically plausible pathophysological mechanism should explain how GERD can cause CRS.
3. clinical manifestations of the suspected GERD-related CRS should respond to anti-reflux therapy.

There are Some theories for the relation between gastric reflux and CRS. The first one is the direct exposure of the nasal and nasopharyngeal mucosa to gastric acid causing inflammation of the mucosa and impaired mucociliary clearance which could cause obstruction of sinus ostia and recurrent infections. It is known that pH variations affect ciliary motility and morphology in the respiratory mucosa.The second hypothesis is a relationship mediated by the vagus nerve; a mechanism already proven in the lower airway and in the nasal mucosa of patients with rhinitis but not in patients with CRS.

Dysfunction of the autonomic nervous system can lead to reflex sinonasal swelling and inflammation, and consequent blockage of the ostia. Demonstrated that by infusing saline with hydrochloric acid in the lower esophagus of healthy volunteers, there was increased production of nasal mucus, increased score of nasal symptoms, and reduced peak nasal inspiratory flow.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged from18-50 years who have been diagnosed to have gastric reflux by gastroenterology departement before the start of treatment, and they also have sinonasal symptoms.

Exclusion Criteria:

* Pregnant
* Significant nasal cavity malformations
* Oncological pathology
* Other sinonasal diseases

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient aged from18-50 years who have been diagnosed to have gastric reflux by gastroenterology departement before the start of treatment, and they also have sinonasal symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
study of correlation between sinonasal troubles & GERD | baseline
  patients diagnosed with GERD who complain of sinonasal symptoms will evaluated for their response after 2 months trial of medical treatment for GERD

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Shaker, Study Chair — Assiut University; Mahmoud Ali, Study Director — Assiut University

REFERENCES:
- [Background] Peery AF, Dellon ES, Lund J, Crockett SD, McGowan CE, Bulsiewicz WJ, Gangarosa LM, Thiny MT, Stizenberg K, Morgan DR, Ringel Y, Kim HP, DiBonaventura MD, Carroll CF, Allen JK, Cook SF, Sandler RS, Kappelman MD, Shaheen NJ. Burden of gastrointestinal disease in the United States: 2012 update. Gastroenterology. 2012 Nov;143(5):1179-1187.e3. doi: 10.1053/j.gastro.2012.08.002. Epub 2012 Aug 8. PMID 22885331
- [Background] Vakil N, van Zanten SV, Kahrilas P, Dent J, Jones R; Global Consensus Group. The Montreal definition and classification of gastroesophageal reflux disease: a global evidence-based consensus. Am J Gastroenterol. 2006 Aug;101(8):1900-20; quiz 1943. doi: 10.1111/j.1572-0241.2006.00630.x. PMID 16928254
- [Background] Vaezi MF, Katzka D, Zerbib F. Extraesophageal Symptoms and Diseases Attributed to GERD: Where is the Pendulum Swinging Now? Clin Gastroenterol Hepatol. 2018 Jul;16(7):1018-1029. doi: 10.1016/j.cgh.2018.02.001. Epub 2018 Feb 7. PMID 29427733
- [Background] Herbella FA, Patti MG. Gastroesophageal reflux disease: From pathophysiology to treatment. World J Gastroenterol. 2010 Aug 14;16(30):3745-9. doi: 10.3748/wjg.v16.i30.3745. PMID 20698035
- [Background] Tasker A, Dettmar PW, Panetti M, Koufman JA, P Birchall J, Pearson JP. Is gastric reflux a cause of otitis media with effusion in children? Laryngoscope. 2002 Nov;112(11):1930-4. doi: 10.1097/00005537-200211000-00004. PMID 12439157
- [Background] O'Reilly RC, He Z, Bloedon E, Papsin B, Lundy L, Bolling L, Soundar S, Cook S, Reilly JS, Schmidt R, Deutsch ES, Barth P, Mehta DI. The role of extraesophageal reflux in otitis media in infants and children. Laryngoscope. 2008 Jul;118(7 Part 2 Suppl 116):1-9. doi: 10.1097/MLG.0b013e31817924a3. PMID 18594333
- [Background] Green BT, Broughton WA, O'Connor JB. Marked improvement in nocturnal gastroesophageal reflux in a large cohort of patients with obstructive sleep apnea treated with continuous positive airway pressure. Arch Intern Med. 2003 Jan 13;163(1):41-5. doi: 10.1001/archinte.163.1.41. PMID 12523915
- [Background] Loehrl TA, Smith TL, Darling RJ, Torrico L, Prieto TE, Shaker R, Toohill RJ, Jaradeh SS. Autonomic dysfunction, vasomotor rhinitis, and extraesophageal manifestations of gastroesophageal reflux. Otolaryngol Head Neck Surg. 2002 Apr;126(4):382-7. doi: 10.1067/mhn.2002.123857. PMID 11997777
- [Background] Holma B, Lindegren M, Andersen JM. pH effects on ciliomotility and morphology of respiratory mucosa. Arch Environ Health. 1977 Sep-Oct;32(5):216-26. doi: 10.1080/00039896.1977.10667285. PMID 20855
- [Background] Lodi U, Harding SM, Coghlan HC, Guzzo MR, Walker LH. Autonomic regulation in asthmatics with gastroesophageal reflux. Chest. 1997 Jan;111(1):65-70. doi: 10.1378/chest.111.1.65. PMID 8995994
- [Background] Wong IW, Rees G, Greiff L, Myers JC, Jamieson GG, Wormald PJ. Gastroesophageal reflux disease and chronic sinusitis: in search of an esophageal-nasal reflex. Am J Rhinol Allergy. 2010 Jul-Aug;24(4):255-9. doi: 10.2500/ajra.2010.24.3490. PMID 20819461
- [Background] Harding SM, Richter JE. The role of gastroesophageal reflux in chronic cough and asthma. Chest. 1997 May;111(5):1389-402. doi: 10.1378/chest.111.5.1389. No abstract available. PMID 9149599
- [Background] Fokkens WJ, Lund VJ, Mullol J, Bachert C, Alobid I, Baroody F, Cohen N, Cervin A, Douglas R, Gevaert P, Georgalas C, Goossens H, Harvey R, Hellings P, Hopkins C, Jones N, Joos G, Kalogjera L, Kern B, Kowalski M, Price D, Riechelmann H, Schlosser R, Senior B, Thomas M, Toskala E, Voegels R, Wang de Y, Wormald PJ. EPOS 2012: European position paper on rhinosinusitis and nasal polyps 2012. A summary for otorhinolaryngologists. Rhinology. 2012 Mar;50(1):1-12. doi: 10.4193/Rhino12.000. PMID 22469599
- [Background] Belafsky PC, Postma GN, Koufman JA. Validity and reliability of the reflux symptom index (RSI). J Voice. 2002 Jun;16(2):274-7. doi: 10.1016/s0892-1997(02)00097-8. PMID 12150380